CLINICAL TRIAL: NCT06738719
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Phase 3 Study to Evaluate the Efficacy and Safety of Subcutaneous CT-P13 in Patients With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: A Phase 3 Study to Evaluate Efficacy & Safety of Subcutaneous CT-P13 in Patients With Moderate to Severe Active Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P13 3.11
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Moderately to Severely Active Rheumatoid Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT-P13 Auto-Injector (Experimental): CT-P13 SC(Subcutaneous) Auto-Injector
  Interventions: Biological: CT-P13 SC Auto-Injector
- Placebo Auto-Injector (Placebo Comparator): Placebo Auto-Injector
  Interventions: Biological: Placebo Auto-Injector

INTERVENTIONS:
Biological: CT-P13 SC Auto-Injector — Subcutaneous(SC) Injection
  Arms: CT-P13 Auto-Injector
Biological: Placebo Auto-Injector — Subcutaneous(SC) Injection
  Arms: Placebo Auto-Injector

SUMMARY:
This is a Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Phase 3 Study to Evaluate the Efficacy and Safety of Subcutaneous CT-P13 in Patients with Moderately to Severely Active Rheumatoid Arthritis

ELIGIBILITY:
[Main Inclusion Criteria]

1. Patient who is male or female aged 18 to 75 years old (both inclusive).
2. Patient who has a diagnosis of RA at least 24 weeks prior to the first administration of the study drug (Day 1) and fulfill the 2010 ACR/EULAR classification criteria for RA.
3. Patient who has active disease as defined by the presence of 6 or more swollen joints (of 66 assessed), 6 or more tender joints (of 68 assessed), and either a high-sensitivity C-reactive protein (hsCRP) ≥1.0 mg/dL (≥10 mg/L) or an erythrocyte sedimentation rate (ESR) ≥28 mm/hour at Screening.
4. Patient who has been receiving the treatment of oral or parenteral dosing with MTX for at least 12 weeks and has been on stable dosing with MTX between 10 to 25 mg/week for at least 4 weeks prior to the first administration of the study drug (Day 1).
5. Patient who has adequate renal and hepatic function at Screening

[Main Exclusion Criteria]

1. Patient who has previously received investigational or licensed product; biological agents or targeted synthetic disease-modifying antirheumatic drugs (DMARDs) (e.g., tofacitinib, baricitinib) for the treatment of RA and/or a tumor necrosis factor (TNF) α inhibitors for the any purpose.
2. Patient who has allergies to any of the excipients of infliximab or any other murine and/or human proteins or patient with a hypersensitivity to immunoglobulin product.
3. Patient who has received or has plan to receive any of prohibited medications or treatments as defined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving clinical response according to the ACR20 criteria at Week 12 | Week 0 ~ Week 12
  To demonstrate superiority of CT P13 SC over Placebo in terms of efficacy as determined by clinical response according to the American College of Rheumatology (ACR) definition of a 20% improvement (ACR20) at Week 12

SECONDARY OUTCOMES:
Change from baseline in HAQ-DI at Week 12 | Week 0 ~ Week 12
  Difference in mean change from baseline in HAQ-DI between treatment groups (CT-P13 SC and Placebo)
Evaluate Pharmacokinetics of CT-P13 SC | Up to 52 Weeks
  Serum concentration of infliximab
Evaluate Safety of CT-P13 SC | Up to 52 Weeks
  * Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
  * All reported terms of AEs will be coded to system organ class (SOC) and preferred term (PT) according to the Medical Dictionary for Regulatory Activities (MedDRA) and severity grading of AEs will be recorded according to the CTCAE Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Klinika Reuma Park Sp. z.o.o, Warsaw, Poland